CLINICAL TRIAL: NCT05609188
Title: Increasing Financial and Health Equity Among Low Income Black Youth and Young Adults
Brief Title: Black Economic Equity Movement
Acronym: BEEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Oregon Health and Science University (Other); MyPath (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1U01OD033266-01 (NIH); 1U01OD033266-01 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Wellness 1; Health Care Utilization; Financial Hardship; Education, Professional
MeSH Terms: conditions — Patient Acceptance of Health Care; Financial Stress

STUDY DESIGN:
Intervention Model Description: The BEEM project is a randomized controlled crossover trial in which 300 low-income Black Emerging Adults (BEA) (aged 18-24) are allocated to receive a $500/month Guaranteed Income (GI) either during the first twelve months of follow-up (phase I) or to receive GI in the second 12 months of a total of 24 months follow-up (phase II). Throughout the study all participants will be offered enrollment in financial capability programs (i.e., peer learning circles and financial coaching) to bolster GI effectiveness.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking the study personnel to randomization group is not possible given that staff need to discuss the randomization with participants upon enrollment. Staff responsible for the financial capability services can not be masked to randomization arm as the participants are free to discuss their experience in the program, including whether and when they are receiving payments.
  The investigators and the senior biostatistician running the final model will be masked to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cash now (Experimental): Participants allocated to the "cash now" arm will receive a $500/month Guaranteed Income (GI) during the first twelve months of follow-up (Phase 1) and no GI in the second twelve months of follow-up (Phase 2).
  Interventions: Other: Guaranteed Income; Behavioral: Peer learning circles; Behavioral: Financial coaching
- Cash in a year (Other): Participants allocated to the "cash in a year" arm will receive no Guaranteed Income (GI) during the first twelve months of follow-up (Phase 1) but will receive a $500/month GI in the second twelve months of follow-up (Phase 2).
  Interventions: Other: Guaranteed Income; Behavioral: Peer learning circles; Behavioral: Financial coaching

INTERVENTIONS:
Other: Guaranteed Income — Monthly cash transfer of $500 per month for 12 months.
Behavioral: Peer learning circles — Participants can opt-in to attend peer learning circles (also called My Money Hour), which are discussion groups of 10-12 participants about financial topics co-led by a peer (Black youth) with experience in financial programming and an adult financial coach. My Money Hour sessions will be offered on-line multiple times throughout every month of the project, with rotating themes, to ensure that the 50-minute sessions are available different days of the week and times of the day.
Behavioral: Financial coaching — Participants can opt-in to receive financial coaching sessions with a trained financial mentor. Meetings will occur monthly and typically include six one hour sessions. The mentor will be responsive to individual needs, but will touch on the following priority areas: building credit (credit repair, improving credit scores, credit products); savings (emergency savings plans, savings habits and strategies, understanding savings accounts); money management (creating budgets, understanding income vs expense, assessing spending, making better financial decisions); financial products (credit building products, auto loans, credit cards); and long-term goals (home ownership, investments).

SUMMARY:
The primary goal is to understand the potential impacts of Guaranteed Income (GI) on Black youth and young adults' financial, emotional, and physical well-being. The main question it aims to answer is: What are the impacts of GI on Black young adults' investments in their future, mental health and unmet mental and sexual/reproductive health service needs? Participants will receive guaranteed income for 12 months and will be offered enrollment in financial capability programs.

DETAILED DESCRIPTION:
The BEEM project is a randomized controlled crossover trial in which 300 low-income Black Emerging Adults (BEA) (aged 18-24) are allocated to receive a $500/month Guaranteed Income (GI) either during the first twelve months of follow-up (phase I) or to receive GI in the second 12 months of a total of 24 months follow-up (phase II). All participants will be offered enrollment in financial capability programs (including peer learning circles and individual financial coaching) to bolster GI effectiveness and will also receive a periodic cell phone-based text messages to ensure that BEA with unmet health service needs receive referrals. The investigators hypothesize that this intervention will increase BEA's investment in their future (education, employment training), improve mental health (depression, anxiety), and reduce unmet mental health and sexual/reproductive health service needs.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-24 years of age at enrollment
* Self-Identify as African American or Black
* Live in a low-income housing tax credit (LIHTC) qualified census tract (QCT) in San Francisco or Oakland. Youth who are homeless or marginally housed in San Francisco and Oakland are also eligible; those who are marginally housed will need a letter from a youth agency that can affirm their marginal housing status.
* Must not be currently enrolled in another GI project
* Must have lived in the US for at least 3 years.
* Must provide informed consent

Exclusion Criteria:

* Participation in another GI program at the time of enrollment
* Lived in the United States for less than 3 years
* Have plans to permanently leave the Bay Area
* Being under the influence of alcohol or other substances at the time of enrollment.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with a Possible Major, Probable Major, or Major Depressive Episode | 12 months of follow-up
  Using the Center for Epidemiologic Studies Depression Scale Revised (CESDR-10), a 'major depressive episode' is defined as 1) presence of anhedonia (inability to feel pleasure), dysphoria (generalized dissatisfaction with life), or irritability 'all the time' or 5-7 days for the past week and 2) at least 4 additional symptoms occurring 'all the time' or 5-7 days in the past week. A 'probable major depressive episode' is defined as 1) presence of anhedonia, dysphoria or irritability nearly every day for the past week, and 2) an additional 3 symptoms occurring 'all the time' or 5-7 days in the past week. A 'possible major depressive episode' is defined as 1) presence of anhedonia, dysphoria or irritability nearly every day for the past week, and 2) an additional 2 symptoms occurring 5-7 days in the past week. The analysis plan includes use of repeated measures to estimate the difference in depressive symptoms at 12 months between study arms relative to baseline proportion.
Proportion of Participants Reporting Investments in the future | 12 months of follow-up
  Indication of enrollment in education, certification, or employment training programs. The analysis plan includes use of repeated measures to estimate the difference in investments in the future at 12 months between study arms relative to baseline proportion.
Proportion of Participants with Unmet Mental Health Service Needs | 12 months of follow-up
  Defined as the absence of receiving mental health care when needed. Unmet mental health need will be assessed by possible, probably or major depressive episode per the CESDR-10 or ≥ 10 on the brief Generalized Anxiety Disorder scale (GAD-7), and not reporting that care was utilized. Service utilization is based on self-report as stating "no" to having accessed any MH service from any kind of health professional. The analysis plan includes the use of repeated measures to estimate the difference in unmet mental health service needs between study arms.
Unmet Sexual and Reproductive Health Service Needs | 12 months of follow-up
  Defined as the absence of receiving sexual and reproductive health services when needed, including STI testing and family planning. This will be measured as self-reported need for SRH (having symptoms of an STI, unprotected sex, or being at risk of unwanted pregnancy) and not reporting that SRH services were utilized. Service utilization is based on self-report as stating "no" to having accessed any SRH service from any kind of health professional. The analysis plan includes the use of repeated measures to estimate the difference in unmet sexual and reproductive health service needs between study arms.

SECONDARY OUTCOMES:
Savings: Proportion of participants with saving to cover a $400 expense | Baseline and 12 months
  Participants will self-report having enough savings to cover an unexpected expense of $400.
Proportion of Participants with Debt | Baseline and 12 months
  Self- reported holding of debt, including: fraudulent debt, owed child support, banking/overdraft fees, bail debts, school debts, utility debts, and credit card or payday loan debt.
Credit score | Baseline and 12 months
  Having a good credit score, defined as a FICO score of 680 points or higher vs. no credit (being credit invisible) or having low a credit score, defined as a FICO score of less than 680.
Proportion of participants with Generalized Anxiety | 12 months of follow-up
  Score of 10 or above on the brief Generalized Anxiety Disorder scale (GAD-7) represents moderate to severe anxiety. The GAD-7 scale ranges from 0-21 with higher scores indicating more generalized anxiety. The analysis plan includes the use of repeated measures to estimate the difference in generalized anxiety at 12 months between study arms relative to baseline proportion.
Hope for the future | Baseline and 12 months
  Hope will be measured using the Hope Matters scale, including 12 items that elicit future expectancy characterized by an individual's perception that a desirable future outcome can be achieved. Participants' level of hope will be classified by using a mean score, with a range of 1-4, with increasing values signifying higher levels of hope.
Financial Capability Score | Baseline and 12 months
  A composite measure of financial knowledge, skills, practices, and mindset

CONTACTS AND LOCATIONS:
Overall Officials: Sheri A Lippman, PhD, Principal Investigator — University of California, San Francisco; Marguerita Lightfoot, PhD, Principal Investigator — Oregon Health & Science University-Portland State University School of Public Health; Margaret Libby, MSW, Principal Investigator — MyPath
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Lippman SA, Libby MK, Nakphong MK, Arons A, Balanoff M, Mocello AR, Arnold EA, Shade SB, Qurashi F, Downing A, Moore A, Dow WH, Lightfoot MA. A guaranteed income intervention to improve the health and financial well-being of low-income black emerging adults: study protocol for the Black Economic Equity Movement randomized controlled crossover trial. Front Public Health. 2023 Nov 3;11:1271194. doi: 10.3389/fpubh.2023.1271194. eCollection 2023. PMID 38026401
- See also: Project website — https://beemproject.org/